CLINICAL TRIAL: NCT04866992
Title: Prospective Registry Trial for Single Port Robot-assisted Nipple Sparing Mastectomy
Brief Title: Prospective Registry Trial for Single Port Robot-assisted Nipple Sparing Mastectomy (SPrNSM)
Acronym: SPrNSM
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Deborah Farr, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU-2019-0522
Record Dates: First submitted 2021-04-01; First posted 2021-04-30 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Ductal Carcinoma in Situ; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; BRCA1 Mutation; BRCA2 Mutation
Keywords: Nipple Sparing Mastectomy; Robot-assisted Nipple Sparing Mastectomy
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a prospective registry trial to determine the outcomes of single port robot-assisted nipple sparing mastectomy (SPrNSM) utilitzing the SP da Vinci surgical system.

DETAILED DESCRIPTION:
Robotic assisted nipple sparing mastectomies with multi-port robots, like the Da Vinci Xi, have been described previously but pose significant hurdles due to the small area like the breast. The Single-Port da Vinci SP (Intuitive Surgical), which was designed for application to small cavity surgery, may be more appropriately suited for this procedure. This is a prospective registry trial to study the outcomes of performing a single-port robot-assisted nipple sparing mastectomy.

Subjects who undergo rNSM and bilateral breast reconstruction of the affected breast via single site small hidden axillary scar technique will be offered participation in the prospective registry trial at their pre-operative visit in the UT Southwestern Breast Clinic. The patient will then be seen at their regularly scheduled clinic appointments at 2 weeks, 1 month, 6 months, and 1 year post operatively at both Breast and Plastics and Reconstructive Surgery (PRS) departments. Outcomes will be tracked in a prospectively kept electronic registry.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age >= 18 years who undergo robotic nipple sparing mastectomy and breast reconstruction with prosthesis at UTSW

Exclusion Criteria:

1. Subjects who are <18 years of age
2. Subjects who do not undergo robotic nipple sparing mastectomy and breast reconstruction with prosthesis at UTSW

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult women who undergo robotic nipple sparing mastectomy (rNSM) with reconstruction.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Feasibility of completion of SPrNSM through axillary incision | Up to 1 year
  Measure number of patients who completed surgery with en bloc removal of the breast through axillary incision v. conversion to open incision
Complication rate of patients requiring re-operation | Up to 1 year
  Number of patients with bleeding requiring a second surgery after SPrNSM
Complication rate of patients with infection requiring explantation of tissue expander | Up to 1 year
  Number of patients with infection after surgery requiring explantation of tissue expander
Complication rate of patients with mastectomy flap necrosis | Up to 1 year
  number of patients with skin, or nipple-areolar flap necrosis using SKIN flap score
Operative surgery time trends with peri-operative outcomes | Up to 1 year
  Measure total surgery time in relation to other outcomes in each patient

SECONDARY OUTCOMES:
Patient reported outcomes | Up to 1 year
  Patient satisfaction is measured using BREAST-Q. Possible scores range from 1-10 Likert scale, with higher scores indicating better/ worse outcome.
Patient reported outcomes | Up to 1 year
  Skin and nipple sensation post operatively with Semmes Weinstein monofilament exam

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Farr, M.D., Principal Investigator — UT Southwestern
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
The study share data of individual participants.